CLINICAL TRIAL: NCT03311958
Title: Molecular Monitoring With Circulating Tumor DNA and Nivolumab Maintenance: A Pilot Study in Diffuse Large B-Cell Lymphoma
Brief Title: Molecular Monitoring With Circulating Tumor DNA and Nivolumab Maintenance
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-110
Record Dates: First submitted 2017-10-05; First posted 2017-10-17 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Regular testing of DLBCL patients who have successfully undergone chemotherapy and are negative for ctDNA. Treatment of patients who become positive for ctDNA with Nivolumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental)
  Interventions: Drug: Nivolumab, IV, 240 mg

INTERVENTIONS:
Drug: Nivolumab, IV, 240 mg — Patients would be given an infusion of 240 mg nivolumab over 30 min

SUMMARY:
Patients suffering from diffuse large B-cell lymphoma (DLBCL) who relapse within 12 months of chemotherapy usually undergo salvage therapies, followed by autologous transplant with a low success rate. These treatments for relapse have significant toxicities and may not be tolerated well by the patients. These patients need an effective means of identifying relapse at an early time point to be treated effectively. Detection of circulating tumor DNA (ctDNA) has been reported to be a sensitive and more specific method to detect relapse at an early stage compared to PET/ CT scans. Purpose of this trial is to monitor patients who have undergone successful chemotherapy for the presence of ctDNA. Patients who test positive for ctDNA would be treated with Nivolumab for a period of 2 years to avoid complete relapse.

DETAILED DESCRIPTION:
Primary Objective:

To determine if nivolumab administration, as a maintenance strategy in DLBCL patients with high risk of relapse, can convert positive ctDNA to negative ctDNA and/or result in relapse free survival (RFS-ctDNA) of 9 months or longer after positive ctDNA was documented.

Secondary Objectives:

1. To evaluate safety of nivolumab as maintenance drug in post-induction, post-salvage and post-autologous transplant setting
2. Relapse free survival (RFS-ctDNA) for nivolumab treated patients
3. Proportion of patients who are able to convert from ctDNA positive to ctDNA negative after nivolumab treatment
4. To validate NeoLabs assay platform by comparing the results to Clonoseq platform.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a tissue diagnosis of diffuse large B cell lymphoma, with a negative PET/CT scan performed within 28 days of study enrollment, with one of the following clinical features: high risk IPI, ABC-subtype DLBCL, Double hit/ triple hit DLBCL, Ki67>90%, or MYC translocation.
* Patients can have any number of prior therapies and any amount of time period from the last therapy as long as they have complete response as seen in PET/CT at the time of enrolment.
* Patients with prior salvage chemo-immunotherapy, radiation therapy, autologous transplantation are included
* Prior radiation therapy must be completed at least 2 weeks prior to study enrollment
* Autologous transplant must have been done 100 days prior to the study enrollment
* Age > 18 years.
* ECOG performance status ≤ 2
* Life expectancy of at least 3 months
* A formalin fixed tissue block or equivalent of 24 slides of the tumor sample for analyses by Adaptive Sequenta and NeoGenomics must be available for analysis.
* Patients must be off cancer-directed therapy for at least 3 weeks (2 weeks for oral agents prior to day 1 of the study
* Patients must have suitable organ and marrow function as defined below

  * Absolute neutrophil count > 500/mm3
  * Platelets > 20,000/mm3
  * Total bilirubin < 2.5 times the ULN
  * AST/ALT (SGOT/SGPT) < 2 times institutional normal limits
  * Creatinine ≤1.5 times normal institutional limits OR
  * Creatinine clearance > 40 ml/min for patients
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document
* WOCBP and sexually active, non-sterile men must be willing to use acceptable method of contraception. WOCBP must agree to not get pregnant and sexually active, non-sterile men must agree not to impregnate a woman for at least 18 weeks after the last dose of nivolumab

Exclusion Criteria:

* Patients with second malignancies (except monoclonal B cells of undetermined significance, antecendant indolent non Hodgkin lymphoma, non-melanomatous skin cancers, papillary thyroid carcinomas, ductal carcinoma in-situ, superficial bladder cancer, prostate cancer or in situ cervical cancers) are excluded unless a complete remission was achieved at least 3 years prior to enrollment and no additional therapy is required or anticipated to be required during the treatment.
* Subjects with active autoimmune disease or a syndrome that requires systemic corticosteroids
* Subjects who received non-oncology vaccine therapies for prevention of infectious disease within 4 weeks of study drug administration.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 agent
* Any contraindication to therapy with nivolumab
* Prior allogeneic transplantation
* Known hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Patients with documented cure from HCV infection will be included
* Known uncontrolled human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS). Patients with documented controlled HIV infection (CD4 > 200 and undetectable viral load) will be included.
* Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease.
* History of anaphylactic reaction to monoclonal antibody therapy
* Poor psychiatric risk
* Patients receiving other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast feeding. Refer to section 4.4 for further details

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of the rate of conversion from positive to negative ctDNA in nivolumab treated patients | 2 years
  Regular monitoring of ctDNA positive patients on nivolumab until they become ctDNA negative
Evaluation of the rate of conversion from positive to negative ctDNA in nivolumab treated patients | 2 years
  Regular testing of ctDNA in positive patients on nivoluman until clinical relapse

SECONDARY OUTCOMES:
To evaluate adverse events in patients on nivolumab as maintenance drug in post-induction, post-salvage and post-autologous transplant setting | 2 years
  Safety evaluated by the frequency and grade of adverse events, as defined by NCI CTCAE 4.03 criteria, for patients treated with nivolumab, such as, uveitis, abnormal lab report or intercurrent illness
Relapse free survival (RFS-ctDNA) for nivolumab treated patients | 2 years
  RFS will be calculated from the day of nivolumab administration until clinical disease
Proportion of patients who are able to convert from ctDNA positive to ctDNA negative after nivolumab treatment | 2 years
  Number of patients who are ctDNA positive and treated with nivolumab, turn ctDNA negative
To compare the ctDNA results of Clonoseq and Neolabs platform | 2 years
  The results obtained from the two platforms will be compared for the feasibility of NeoLabs platform for detecting any change in ctDNA numbers in blood

CONTACTS AND LOCATIONS:
Overall Officials: Shazia Nakhoda, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States